CLINICAL TRIAL: NCT05142397
Title: The Dynamic Process of Vaginal Microbiota and Mucosal Immunity After Focused Ultrasound Treatment of Cervical Intraepithelial Neoplasia Patients With Fertility Requirement
Brief Title: The Dynamic Process of VMB and Mucosal Immunity After FUS Treatment of CIN Patients With Fertility Requirement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shufang Chang (Other)
Responsible Party: Sponsor-Investigator, Shufang Chang, professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: shfch2005
Record Dates: First submitted 2021-11-03; First posted 2021-12-02 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical secretions、Vaginal microbiota、HPV genotyping、Thinprep cytologic test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated women: HPV positive，pathology result indicate cervical intraepithelial neoplasia
  Interventions: Procedure: Focused Ultrasound
- Healthy controls: HPV negative, normal cytology

INTERVENTIONS:
Procedure: Focused Ultrasound — Focused ultrasound generates heat effects, mechanical effects and cavitation effects that denature the diseased tissues, facilitate necrosis and allow them to be replaced by surrounding normal healthy tissues.
  Other Names: High-Intensity Focused Ultrasound Ablation
  Groups: Treated women

SUMMARY:
Cervical cancer is the fourth leading cause of cancer death in women worldwide, and cervical intraepithelial neoplasia (CIN) can progress to cervical cancer. Therefore, timely treatment of CIN is critical in preventing the occurrence of cervical cancer. With the implementation and promotion of the World Health Organization's 2030 Global Strategy for the Elimination of Cervical Cancer, an increasing number of women are detecting and treating CIN at an earlier stage. Common treatment methods include ablation treatment and excision treatment, but for women who are planning to have children, the risk of cervical insufficiency and pregnancy complications is greatly increased after excisional treatment, so ablation treatment seems to be a better choice.

DETAILED DESCRIPTION:
Focused ultrasound (FUS) is a new ablation method for the treatment of CIN that has received a lot of attention because of its unique ablation mode (from inside to outside) and lack of smoke, ionizing radiation, and other side effects. Preliminary studies have found that FUS treatment is safe and effective at reversing CIN, with curative effects comparable to traditional ablation and excisional treatments. However, few studies have reported the mechanism of FUS in the treatment of CIN. As a kind of ablation treatment, it is unclear whether FUS, like other ablation treatment mechanisms, stimulates the immune response of the body to promote the reversal of the lesions by in situ necrotic lesions.

There is limited evidence to support the link between FUS, immune response, and CIN. Fu compared the cervical tissues of patients with CIN before and after FUS treatment and found that the expression of p16 and ki-67 decreased while the expression of Fas increased after treatment, indicating that FUS can regulate cell proliferation and apoptosis-related proteins, and promote the recovery of cervical tissues. More recently, Zeng compared the cervical immune microenvironment in patients with CIN before and after FUS treatment. It has shown that FUS treatment increased the expression of ERAP1 in cervical tissue and decreased the level of IgA and IL-10 in cervicovaginal lavage, which indicated that FUS treatment can regulate the cervical immune microenvironment.

The immune response of the body is a dynamic and changing process. Any attempt to infer further on immunological changes before and after treatment require dynamic studies that will explore how FUS ablation of the disease, i.e. CIN, will alter the cervical immune microenvironment. The local immunological indexes produced by FUS treatment of CIN should be a dynamic process, and more time points should be selected to monitor the changes in these immunological indexes. Currently, there are no such studies.

At the same time, a large number of studies suggest that Vaginal Microbiota(VMB) can alter the cervicovaginal immune microenvironment and Lactobacillus spp. depleted and high diversity of VMB is prone to form a pro-inflammatory environment, which in turn promotes the progression of CIN and the occurrence of cervical cancer. Therefore, to further explore the mechanisms of FUS ablation treatment of CIN and clearance of HPV, this interventional study was conducted to dynamically observe the changes in the VMB and mucosal immunity in patients with CIN before and after FUS ablation treatment and to compare with untreated healthy controls. This may also have implications for the persistence and recurrence of lesions.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18-60 years old；
2. patients who had sexual life；
3. patients who had HPV infection;
4. patients who apply to ablation therapy
5. pathological report indicates CIN

Exclusion Criteria:

1. pregnant or lactating women;
2. patients who had cervical treatment ;
3. patients who had genital tract infection ;
4. patients who had chronic diseases, such as allergic diseases ，autoimmune diseases and so on；
5. patients who received antibiotics or pessaries within 14 days of sampling.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We plan to include women with HPV positive, who plan for focused ultrasound ablation treatment for CIN attending the colposcopy clinics at the Second Affiliated Hospital of Chongqing Medical University.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunological indexes | We will get specimens in therapeutic day, after treatment 7-10 days，84-112days and 168-196 days respectively.
  Immunological indexes(IFN-γ、IL-8、IL-10、IL-1β、SIgA) in cervical secretions will be measured by enzyme-linked immunosorbent assay (ELISA).
Anti-microbial peptides | We will get specimens in therapeutic day, after treatment 7-10 days，84-112 days and 168-196 days respectively.
  Anti-microbial peptides levels (hBD-1、SLPI ) in cervical secretions will be measured by enzyme-linked immunosorbent assay (ELISA).
Vaginal microbiota | We will get specimens before therapeutic day, after treatment 84-112 days and 168-196 days respectively.
  We will evaluate vaginal microbiota by bacterial diversity and richness, and Lactobacillus grading.
HPV genotyping | We will get specimens before therapeutic day, after 84-112 days and 168-196 days respectively.
  HPV DNA testing and genotyping
Cytology | We will get specimens before therapeutic day, after treatment 84-112 days and 168-196 days respectively.
  Thinprep cytologic test

SECONDARY OUTCOMES:
Measurement of dimensions of cervix | We will measure the dimensions of cervix before therapeutic day and after treatment 84-112 days respectively.
  Transvaginal ultrasonography is performed to measure the dimensions of cervix.
Antisperm antibody | We will get specimens before therapeutic day, after treatment 84-112 days and 168-196 days respectively.
  Antisperm antibody in cervical secretions will be measured by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Shu F Chang, professor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided